CLINICAL TRIAL: NCT03071224
Title: Phase 1 Evaluation of [18F]MK-6240 PET as an Imaging Marker for Tau Protein in the Brain of Patients With Alzheimer's Disease Compared to Healthy Volunteers
Brief Title: Phase 1 Evaluation of [18F]MK-6240 PET as an Imaging Marker for Tau Protein
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: [18F] MNI-946
Record Dates: First submitted 2017-02-28; First posted 2017-03-06 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2019-09

CONDITIONS: Alzheimer Disease; Healthy Volunteers
Keywords: AD; HV
MeSH Terms: conditions — Alzheimer Disease | interventions — florbetapir

ARMS (1):
- [18F]MNI-946 (Experimental): To evaluate [18F]MK-6240 (also known as [18F]MNI-946) a tau targeted radiopharmaceutical.
  Interventions: Drug: [18F] MNI-946; Drug: [18F]Florbetapir

INTERVENTIONS:
Drug: [18F] MNI-946 — Subjects will undergo PET imaging using [18F]MNI-946, a PET radioligand for imaging tau.
  Other Names: [18F]MK6240
Drug: [18F]Florbetapir — Subjects with Alzheimer's disease will receive a [18F]florbetapir scan to compare distribution of tau in the brain compared to that of [18F]MNI-946.

SUMMARY:
The overall goal of this protocol is to evaluate [18F]MK-6240 (also known as [18F]MNI-946) a tau targeted radiopharmaceutical.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate [18F]MK-6240 (also known as [18F]MNI-946) a tau targeted radiopharmaceutical.

* To measure the dynamic uptake and washout of [18F]MK-6240 in brain using positron emission tomography (PET) in patients with Alzheimer's disease and healthy volunteers.
* To measure blood metabolites of [18F]MK-6240 and perform kinetic modeling to assess its ability to measure tau protein in brain using the tracer plasma concentration or a reference region as indirect input.
* To obtain test/retest reliability of the tracer binding parameters in patients with Alzheimer's disease and healthy volunteers (Cohort 1).
* To acquire safety data following injection of [18F]MK-6240.
* To determine the longitudinal change in tau burden (including SUVR and tau distribution metrics) compared to baseline in AD subjects and in similarly aged HV subjects.
* To evaluate the correlation between the longitudinal change in tau burden and change in clinical, MRI and CSF biomarker measures in AD subjects and in similarly-aged HV subjects.
* To further explore the relationship between tracer metabolism and smoking (Cohort 3).

ELIGIBILITY:
Inclusion Criteria (for all subjects all cohorts):

* Written informed consent must be obtained before any assessment is performed.
* Female subjects must be documented by medical records or physician's note to be either surgically sterile (by means of hysterectomy, bilateral oophorectomy, or tubal ligation) or post-menopausal for at least 1 year or, if they are of child-bearing potential, must commit to use two methods of contraception, one of which is a barrier method for the duration of the study.
* Male subjects and their partners of childbearing potential must commit to the use of two methods of contraception, one of which is a barrier method for male subjects for the study duration.
* Male subjects must not donate sperm for the study duration.
* Willing and able to cooperate with study procedures.

Inclusion criteria for healthy volunteer subjects (all cohorts):

* Males and females aged ≥50 years. Healthy with no clinically relevant finding on physical examination at screening and upon reporting for the [18F]MK-6240 imaging visit.
* No cognitive impairment from neuropsychological battery as judged by the investigator
* Have screening [18F]Florbetapir PET imaging demonstrating no significant amyloid binding based on qualitative (visual read).
* No family history of Alzheimer's disease or neurological disease associated with dementia
* Have a CDR global score=0
* Have an MMSE score ≥28
* Willing and able to cooperate with study procedures.

Inclusion criteria for subjects with a diagnosis of probable Alzheimer's disease (AD) all cohorts:

* Males and females aged 50 to 80 years.
* Have probable Alzheimer's disease dementia, based on the NINCDS/ADRDA and DSM-IV criteria, with mild severity and amnestic presentation
* Have a CDR score ≥ 0.5 at screening
* Have a MMSE score between ≤26 .
* Have screening [18F]Florbetapir or prior (in the last 12 months) amyloid PET imaging demonstrating amyloid binding based on qualitative (visual read).[18F]Florbetapir PET imaging results will be shared with participants and scans may be used by participants for future research use.
* A brain MRI that supports a diagnosis of AD, with no evidence of significant neurologic pathology.
* Medications taken for symptomatic treatment of AD must be maintained on a stable dosage regimen for at least 30 days before screening visit.
* Signed and dated written informed consent obtained from the subject and the subject's legally authorized representative or caregiver (if applicable).
* The subject has an appropriate caregiver capable of accompanying subject on all visits, if necessary.

Inclusion Criteria for all AD and HV subjects in Cohort 3:

• Subjects must be active smokers at the time of initial consent

Exclusion Criteria (for aAll subjects all cohorts):

* Current or prior history of any alcohol or drug abuse.
* Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
* Subject has received an investigational therapeutic drug or device within 30 days of screening.
* Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines.
* Pregnancy, lactating or breastfeeding.
* Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
* Unsuitable veins for repeated venipuncture.
* MRI exclusion criteria include: Findings that may be responsible for the neurologic status of the subject such as significant evidence of cerebrovascular disease (more than two lacunar infarcts, any territorial infarct >1cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the FLAIR sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with CNS disease.
* Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.

Exclusion criteria for subjects with AD ( all cohorts):

• Has received treatment that targeted Aβ or tau within the last 3 months.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2021-06-09 (Actual); Study Completion 2021-06-09 (Actual)

PRIMARY OUTCOMES:
To determine the longitudinal change in tau burden (including SUVR and tau distribution metrics) compared to baseline in AD subjects and in similarly aged HV subjects. | 1 year
  Tracer uptake will be evaluated in regions of interest for analysis of regional [18F]MK-6240 binding/uptake and expressed in SUV by using established methods for normalization for 12 AD and 3 HV subjects in Cohort 1, 8 AD and 2 HV subjects in Cohort 2, and 3 AD and 3 HV subjects in Cohort 3. Target regions of interest in the standard volume of interest (VOI) template, will be used for tracer uptake quantitation of potentially increased binding to tau pathology will correspond in particular to the cortical regions of the brain. Descriptive statistics will be applied to describe the tau deposition by region as measured by [18F]MK-6240.
  Descriptive statistics will be applied to describe the tau deposition by region as measured by [18F]MNI-946.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph. D, Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Info — http://invicro.com/